CLINICAL TRIAL: NCT02458352
Title: Usefulness of Ultra Low Dose Cardiac CT for Coronary Calcium Scoring and for Attenuation Correction of SPECT
Brief Title: Ultra Low Dose CT for CACS and AC of SPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ-2015-0072
Record Dates: First submitted 2015-05-08; First posted 2015-06-01 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard dose CT, Ultra-low dose CT (Other): Standard dose non-contrast enhanced CT (clinically indicated) and Ultra low dose non-contrast enhanced CT (as part of the trial)
  Interventions: Device: Ultra low dose non-contrast enhanced CT; Device: Standard dose non-contrast enhanced CT

INTERVENTIONS:
Device: Ultra low dose non-contrast enhanced CT — Non-contrast enhanced CT for CACS and AC using a novel protocol for ultra low dose radiation dose exposure
Device: Standard dose non-contrast enhanced CT — Clinically indicated non-contrast enhanced CT for CACS and AC according to routine protocol

SUMMARY:
The aim of the study is to compare the CACS obtained from standard dose CT to the CACS obtained from ultra-low-dose scans. Additionally, the usefulness of ultra-low-dose CT for AC of myocardial perfusion SPECT will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for myocardial perfusion SPECT
* Male and Female subjects ≥18 years of age,
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* CACS of 0 after inclusion of 10 patients with CACS 0
* Stents or implanted cardiac devices (valves, pace makers, ICD)
* Coronary artery bypass grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Treyer, PhD, Study Director — University of Zurich
Locations (1):
- Department of Nuclear Medicine, University Hospital Zurich, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose CT, Ultra-low Dose CT: Standard dose and ultra-low dose non-contrast enhanced CT
  Standard dose non-contrast enhanced CT: Clinically indicated non-contrast enhanced CT for CACS and AC according to routine protocol Ultra-low dose non-contrast enhanced CT: Additional scan as part of the trial
Period: Overall Study
Arm/Group | Standard Dose CT, Ultra-low Dose CT
Started | 105
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Dose CT, Ultra-low Dose CT: Standard dose non-contrast enhanced CT
  Standard dose non-contrast enhanced CT: Clinically indicated non-contrast enhanced CT for CACS and AC according to routine protocol
Arm/Group | Standard Dose CT, Ultra-low Dose CT
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Agreement and Correlation of Coronary Artery Calcium Score Obtained From Ultra-low-dose and Standard CT
Description: CAC and BA limits of agreement between coronary artery calcium score obtained from ultra-low-dose and standard CT.
  Coronary artery calcium (CAC) is a measure for quantification of coronary artery calcification based on non-contrast enhanced CT, ranging from 0 (no calcifications) to infinite. It is an arbitrary unit. Increasing CAC means higher amounts of coronary artery calcifications and is associated with worse prognosis.
  Bland-Altman (BA) analysis is a statistical method to compare two modalities or techniques assessing the same measure. Limits of agreement is defined as +/- twice the standard deviation of the differences between the reference method and the new modality/technique. Broader limits of agreement mean less accurate results obtained by the new modality/techniqe, while a 0 BA limit of agreement would theoretically reflect perfect agreement.
Time Frame: 1 days
Population: 2/105 participants were not analyzed due to corrupt datasets.
Measure: Median (Inter-Quartile Range); unit: Agatston score
Groups:
- Standard Dose CT: Standard dose non-contrast enhanced CT
  Standard dose non-contrast enhanced CT: Clinically indicated non-contrast enhanced CT for CACS and AC according to routine protocol
- Ultra-low Dose CT: Ultra low dose non-contrast enhanced CT
  Ultra low dose non-contrast enhanced CT: Non-contrast enhanced CT for CACS and AC using a novel protocol for ultra low dose radiation dose exposure
Arm/Group | Standard Dose CT | Ultra-low Dose CT
Number analyzed (Participants) | 103 | 103
Agatston score | 212 [25 to 901] | 178 [22 to 764]

2. Primary Outcome: Intra-class Correlation Coefficient Between Segmental Relative Tracer Uptake From SPECT Datasets Reconstructed With AC Maps Based on Ultra-Low-Dose and Standard Dose CT
Description: For every patient, the CT images from 120 and 70 kVp-CT scans were used to create CTAC maps which were then used to reconstruct SPECT images, displayed as a 17-segment model polar plot with normalized percent tracer uptake given for every segment. Intra-class correlation was then applied to compare segmental relative tracer uptake. Analysis and the resulting correlation coefficient of 0.987 basically demonstrates interchangeability between the two datasets.
Time Frame: 1 day
Population: 2/105 participants were not analyzed due to corrupt datasets.
Measure: Number; unit: Intraclass correlation coefficient
Arm/Group | Standard Dose CT | Ultra-low Dose CT
Number analyzed (Participants) | 103 | 103
Intraclass correlation coefficient | 1 | 0.987

ADVERSE EVENTS:
Arm/Group | Standard Dose CT | Ultra-low Dose CT
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes